CLINICAL TRIAL: NCT04448886
Title: Saci-IO HR+: Randomized Phase II Study of Sacituzumab Govitecan With or Without Pembrolizumab in Hormone Receptor-positive (HR+) / HER2- Metastatic Breast Cancer (MBC)
Brief Title: Sacituzumab Govitecan +/- Pembrolizumab In HR+ / HER2 - MBC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ana C Garrido-Castro, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Ana C Garrido-Castro, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-153
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Invasive Breast Cancer; Metastatic Breast Cancer; HR-Positive Breast Cancer; HER2-negative Breast Cancer
Keywords: Invasive Breast Cancer; Metastatic Breast Cancer; HR-Positive Breast Cancer; HER2-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sacituzumab Govitecan + Pembrolizumab (Experimental): The research study procedures include: screening for eligibility, research blood collections, at least two research biopsies, paired research stool collections, and study treatment including evaluations and follow up visits. Each Cycle =21 Days
  * Sacituzumab Govitecan (iv) fixed dose, administered twice per cycle
  * Pembrolizumab (iv) fixed dose administered once per cycle
  Interventions: Drug: Pembrolizumab; Drug: Sacituzumab Govitecan
- Sacituzumab Govitecan (Experimental): The research study procedures include: screening for eligibility, research blood collections, at least two research biopsies, paired research stool collections, and study treatment including evaluations and follow up visits.
  - Sacituzumab Govitecan (iv) fixed dose, administered twice per cycle
  Interventions: Drug: Sacituzumab Govitecan
- Retreatment (Experimental): Participants who have attained a confirmed complete response (CR) who have been treated for at least 24 weeks on protocol therapy and had at least three cycles (with pembrolizumab and sacituzumab govitecan (Arm A) or sacituzumab govitecan alone (Arm B)) beyond the date when the initial CR was declared may be eligible for additional sacituzumab govitecan and/or pembrolizumab therapy if they progress after stopping study treatment. This retreatment is termed the Second Course Phase of this study and is only available if the study remains open and the subject meets protocol-specified conditions.
  Interventions: Drug: Pembrolizumab; Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Pembrolizumab — (iv) fixed dose, administered once per cycle
  Other Names: Keytruda
  Arms: Retreatment; Sacituzumab Govitecan + Pembrolizumab
Drug: Sacituzumab Govitecan — (iv) fixed dose, administered twice per cycle
  Other Names: TRODELVY

SUMMARY:
This research study is evaluating the safety and effectiveness of Sacituzumab Govitecan with or without Pembrolizumab in metastatic HR+/HER2- breast cancer.

The names of the study interventions involved in this study are:

* Sacituzumab govitecan (IMMU-132)
* Pembrolizumab (Keytruda®; MK-3475)

DETAILED DESCRIPTION:
The research study procedures include: screening for eligibility, research blood collections, at least two research biopsies, paired research stool collections, and study treatment including evaluations and follow up visits.

The names of the study interventions involved in this study are:

* Sacituzumab govitecan (IMMU-132)
* Pembrolizumab (Keytruda®; MK-3475)
* Questionnaires/Data Collection/Sample Collection

Participants will be randomized into one of two groups. Group A: Sacituzumab govitecan (IMMU-132) and Pembrolizumab Group B: Sacituzumab govitecan (IMMU-132)

Participants will receive study treatment for as long they are benefiting from the therapy. Participants will be followed for the rest of their lives. It is expected that about 110 people will take part in this research study

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug or a combination of investigational drugs to learn whether the drug or drug combination works in treating a specific disease. "Investigational" means that the drug or drug combination is being studied. The U.S. Food and Drug Administration (FDA) has not approved Sacituzumab Govitecan for your specific disease, but it has been approved for other uses. The U.S. Food and Drug Administration (FDA) has not approved Pembrolizumab for your specific disease but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer with unresectable locally advanced or metastatic disease. Participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation, i.e. visible chest wall disease or metastases on imaging meeting standard radiology criteria (i.e. lymph nodes larger than 1 cm in the short axis diameter).
* Participants must have HR-positive, HER2-negative breast cancer (ER>1% and/or, PR>1%, HER2-negative per ASCO CAP guidelines) on local pathology review. If a patient has more than one histological result, the most recent sample will be considered for inclusion.
* Participants must have either progressed on or within 12 months of adjuvant endocrine therapy or have progressed on at least one line of endocrine therapy for metastatic disease, and be considered appropriate candidates for chemotherapy.
* Participants must have evaluable or measurable disease per RECIST 1.1. For instance, patients with bone only disease will be allowed to participate.
* Participants must agree to undergo a research biopsy, if tumor is safely accessible, at baseline. Previously collected archival tissue will also be obtained on all participants. Tissue needs to be located and availability confirmed at time of registration. Participants must agree to a mandatory repeat biopsy 3-6 weeks after starting treatment, if tumor is safely accessible.
* Prior chemotherapy: Participants may have received 0-1 prior chemotherapeutic regimens for metastatic breast cancer and must have been off treatment with chemotherapy for at least 14 days prior to study treatment initiation. If a prior chemotherapy was given for less than 1 cycle, it will not be counted as a prior line. No prior irinotecan or topoisomerase I-containing antibody drug conjugates in the metastatic or neo/adjuvant setting are allowed. All toxicities related to prior chemotherapy must have resolved to CTCAE v5.0 grade 1 or lower, except alopecia can be any grade and neuropathy can be grade 2 or lower.
* Prior biologic therapy: Patients must have discontinued all biologic therapy at least 14 days prior to study treatment initiation. All toxicities related to prior biologic therapy must have resolved to CTCAE v5.0 grade 1 or lower.
* Prior targeted therapy: Targeted therapy must have been discontinued ≥ 14 days prior to initiation of study therapy. All toxicities related to prior targeted therapy must have resolved to CTCAE v5.0 grade 1 or lower.
* Prior radiation therapy: Patients may have received prior radiation therapy. Radiation therapy must be completed at least 7 days prior to the initiation of study treatment (at least 7 days for SRS), and all toxicities related to prior radiation therapy must have resolved to CTCAE v5.0 grade 1 or lower, unless otherwise specified per protocol. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Previously treated brain metastases are permitted, with the following provisions:

  * Prior SRS should complete ≥ 7 days before study treatment initiation
  * Prior WBRT should complete ≥ 7 days before study treatment initiation.
  * Any corticosteroid use for brain metastases must have been discontinued for ≥ 7 days prior to study treatment initiation.
* Participants on bisphosphonates or RANK ligand inhibitors may continue receiving therapy during study treatment and also may initiate therapy with these agents on study if clinically indicated.
* The subject is ≥ 18 years old.
* ECOG performance status 0-1 (Karnofsky > 60%).
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,000/mcL
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥ 9.0 g/dl
  * INR/PT/aPTT ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is in therapeutic range of anticoagulant
  * Total bilirubin ≤1.5 × institutional upper limit of normal (ULN) (or ≤2.0 x ULN in patients with documented Gilbert's Syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN or ≤5 × institutional ULN for participants with documented liver metastases
  * Serum creatinine ≤1.5 × institutional ULN OR creatinine clearance ≥ 30 mL/min/ 1.73m2 for participants with creatinine levels above institutional ULN.
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 2 weeks prior to study treatment initiation. Childbearing potential is defined as participants who have not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and have not undergone surgical sterilization (removal of ovaries and/or uterus).
* Women of childbearing potential (WOCBP) must agree to use an adequate method of contraception. Contraception is required starting with the first dose of study medication through 180 days (6 months) after the last dose of study medication. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, and copper intrauterine devices. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. Hormonal contraceptives are contraindicated for HR+ breast cancer.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with pembrolizumab and 3 months after the last dose of study treatment.
* The participant must be capable of understanding and complying with the protocol and willing to sign a written informed consent document.

Exclusion Criteria:

* Prior therapy with any anti-PD-1, PD-L1, or PD-L2 agent or sacituzumab govitecan. Prior therapy with irinotecan or topoisomerase I-containing antibody drug conjugates at any time for early stage or metastatic disease.
* Prior hypersensitivity to the excipients of pembrolizumab or sacituzumab govitecan therapy.
* Known history of UDP-glucuronosyltransferase 1A1 (UGT1A1) *28 allele homozygosity, which is associated with increased risk for neutropenia and diarrhea related to irinotecan.

Note: Concurrent administration of strong UGT1A1 inhibitors or inducers is not allowed during the course of the study.

* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms.
* Major surgery within 2 weeks prior to study treatment initiation. Patients must have recovered from any effects of any major surgery.
* Uncontrolled, significant intercurrent or recent illness including, but not limited to, ongoing or active infection, uncontrolled non-malignant systemic disease, uncontrolled seizures, or psychiatric illness/social situation that would limit compliance with study requirements in the opinion of the treating investigator.
* Participant has a medical condition that requires chronic systemic steroid therapy (> 10 mg of prednisone daily or equivalent) or any other form of immunosuppressive medication (including disease modifying agents) and has required such therapy in the last 2 years. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic therapy.
* Participant has documented history of autoimmune disease or syndrome that currently requires systemic steroids or immunosuppressive agents.
* History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
* Individuals with a history of a second malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers that have been diagnosed and treated within the past 3 years are eligible: cervical/prostate carcinoma in situ, superficial bladder cancer, non-melanoma cancer of the skin. Patients with other cancers diagnosed within the past 3 years and felt to be at low risk of recurrence should be discussed with the study principal investigator to determine eligibility.
* Participant has a known history of human immunodeficiency virus (HIV), Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as detected HCV RNA [qualitative]) infection. HIV-positive participants are ineligible due to the potential for pharmacokinetic interactions of combination antiretroviral therapy with study drugs and the increased risk of fatal infections. Note: No testing for HIV, Hepatitis B, or Hepatitis C is required unless mandated by local health authority.
* The participant has received a live vaccine within 28 days prior to study treatment initiation. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. The use of the inactivated seasonal influenza vaccine is allowed.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* It is unknown whether pembrolizumab is excreted in human milk. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, participants who are breast-feeding are not eligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2027-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Garrido-Castro, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - DFCI @ Foxborough, Foxborough, Massachusetts
  - DFCI @ Milford Regional Hospital, Milford, Massachusetts
  - DF/BWCC in Clinical Affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Pennsylvania-Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: https://www.dana-farber.org/research/innovations

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated in September 2020 and closed accrual in January 2024. Patients were enrolled from the following sites: University of Chicago, DFCI (Boston, Milford, South Shore, Foxborough), Emory University, University of Pennsylvania, and University of North Carolina (Chapel Hill).
Pre-assignment Details: Prior to amendment 3 of the study protocol, the enrolled patient were initially entered into prescreen phase, to verify that their PD-L1+ was greater or equal to 10 by centrally tested 22C3 combined positive score prior to proceeding for the study. This restriction was lifted starting from amendment 3.
Period: Overall Study
Arm/Group | Sacituzumab Govitecan + Pembrolizumab | Sacituzumab Govitecan
Started | 52 | 52
Completed | 48 | 51
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Population: A total of 110 patients were randomized. However, 6 out of 110 patients did not start treatment (4 did not meet eligibility, 1 withdrew consent prior to starting treatment, 1 died prior to starting treatment). Therefore a total of 104 patients that started treatment were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sacituzumab Govitecan + Pembrolizumab | Sacituzumab Govitecan | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Median (Full Range); unit: Year] | 56.5 [31 to 81] | 57 [27 to 80] | 57 [27 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 102
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 40 | 44 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 46 | 49 | 95
  Unknown or Not Reported | 4 | 1 | 5
ER status at closest date prior to enrollment [Count of Participants; unit: Participants]
  Positive (>=1% cell staining) | 52 | 52 | 104
  Negative (<1% cell staining) | 0 | 0 | 0
PR status at closest date prior to enrollment [Count of Participants; unit: Participants]
  Positive (>=1% cell staining) | 25 | 27 | 52
  Negative (<1% cell staining) | 27 | 25 | 52
Prior lines of chemotherapy for primary tumor [Count of Participants; unit: Participants]
  Yes | 28 | 28 | 56
  No | 13 | 11 | 24
  N/A | 11 | 13 | 24
Prior lines of chemotherapy for metastatic tumor [Count of Participants; unit: Participants]
  0 line | 26 | 25 | 51
  1 line | 26 | 27 | 53
Prior CDK 4/6 inhibitor for primary tumor [Count of Participants; unit: Participants]
  Yes | 7 | 11 | 18
  No | 34 | 28 | 62
  N/A | 11 | 13 | 24
Prior CDK 4/6 inhibitor for metastatic tumor [Count of Participants; unit: Participants]
  Yes | 46 | 44 | 90
  No | 6 | 8 | 14
Prior CDK 4/6 inhibitor ever (for primary or metastatic) [Count of Participants; unit: Participants]
  Yes | 49 | 48 | 97
  No | 3 | 4 | 7
Endocrine therapy for primary tumor [Count of Participants; unit: Participants]
  Yes | 37 | 39 | 76
  No | 4 | 0 | 4
  N/A | 11 | 13 | 24
Brain metastasis present at enrollment/diagnosis [Count of Participants; unit: Participants]
  Yes | 4 | 5 | 9
  No | 48 | 47 | 95
Liver metastasis present at enrollment/diagnosis [Count of Participants; unit: Participants]
  Yes | 40 | 41 | 81
  No | 12 | 11 | 23
Presentation at metastatic diagnosis [Count of Participants; unit: Participants]
  De novo MBC | 11 | 13 | 24
  Recurrent MBC | 41 | 39 | 80
ECOG PS at enrollment [Count of Participants; unit: Participants] — ECOG performance status criteria = 0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  1: Have symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (ex. light housework, office work)
  Participants
    0 | 38 | 31 | 69
    1 | 14 | 21 | 35

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Compare the progression-free survival (PFS) of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone. PFS is defined as the time from study randomization to disease progression, according to RECIST 1.1 or medical judgment, the latter based on established clinical parameters, such as rising tumor markers and physical exam evidence of progression, i.e. worsening chest wall disease, or death due to any cause, whichever occurred first. Patients alive without disease progression are censored at the date of last disease evaluation.
Time Frame: Assessed at baseline and every 3 cycles/9 weeks with a window of -7 days to + 3 days (e.g., between Cycle 3 Day 15 and Cycle 4 Day 4). Expected study duration to primary analysis of PFS is 38 months. The reported data is as of data cutoff of 3/9/2024.
Population: as for baseline characteristics
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Sacituzumab Govitecan + Pembrolizumab | Sacituzumab Govitecan
Number analyzed (Participants) | 52 | 52
Months | 8.36 [5.30 to 11.05] | 6.45 [3.95 to 8.32]

2. Secondary Outcome: Objective Response Rate
Description: Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing Overall Response Rate (ORR) by RECIST 1.1
Time Frame: Assessed at baseline and every 3 cycles/9 weeks with a window of -7 days to + 3 days (e.g., between Cycle 3 Day 15 and Cycle 4 Day 4). Expected study duration is 38 months. The reported data is as of data cutoff of 3/9/2024.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sacituzumab Govitecan + Pembrolizumab | Sacituzumab Govitecan
Number analyzed (Participants) | 52 | 52
Participants | 15 | 10

3. Secondary Outcome: Overall Survival
Description: Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing overall survival (OS), defined as the time from randomization (or registration) to death due to any cause with censoring at date last known alive, will be reported with Kaplan Meier estimates
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sacituzumab Govitecan + Pembrolizumab | Sacituzumab Govitecan
Number analyzed (Participants) | 52 | 52
Months | 20.0 [16.9 to NA] — We don't have enough number of events to reliably estimate the upper CI | 18.0 [17.1 to 20.0]

4. Secondary Outcome: Clinical Benefit Rate
Description: Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing clinical benefit rate (CBR). CBR defined as CR, PR or stable disease for ≥ 24 weeks according to RECIST 1.1
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sacituzumab Govitecan + Pembrolizumab | Sacituzumab Govitecan
Number analyzed (Participants) | 52 | 52
Participants | 26 | 26

5. Secondary Outcome: Time to Progression
Description: Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing time to progression
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sacituzumab Govitecan + Pembrolizumab | Sacituzumab Govitecan
Number analyzed (Participants) | 52 | 52
Months | 8.36 [5.3 to 12.5] | 6.68 [3.95 to 8.68]

6. Secondary Outcome: Duration of Response
Description: Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing the duration of response (the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or death due to any cause)
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Median (Full Range); unit: Months
Arm/Group | Sacituzumab Govitecan + Pembrolizumab | Sacituzumab Govitecan
Number analyzed (Participants) | 52 | 52
Months | 12.93 [4.14 to NA] — We don't have enough number of events to reliably estimate the upper CI | 4.51 [4.47 to NA] — We don't have enough number of events to reliably estimate the upper CI

ADVERSE EVENTS:
Time Frame: AEs were collected from enrollment to end of treatment (SG was administered until progression; pembrolizumab was administered until progression or a max. of 35 doses (24 months) was reached, whichever occurred first). End of treatment visit (SG +/- pembrolizumab) was to occur within 45 days of final administration of study treatment. Additionally, AE assessment was performed 90 days (-15/+30 days) after the last dose of pembrolizumab. As of 3/9/24 data cutoff, the max. follow-up was 26 months.
Description: For mortality information, all patients that were randomized (n=110) were included as the denominator. For other AE information, only those that started treatment (n=104) are included as the denominator. As of data cutoff of 3/9/2024, the maximum follow-up duration is 26 months.
Arm/Group | Sacituzumab Govitecan + Pembrolizumab | Sacituzumab Govitecan
All-Cause Mortality (participants affected / at risk) | 18/54 | 22/56
Serious Adverse Events (participants affected / at risk) | 40/52 | 36/52
Other Adverse Events (participants affected / at risk) | 49/52 | 48/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan + Pembrolizumab (N=52) | Sacituzumab Govitecan (N=52)
Neutrophil count decreased (Investigations) | 28 | 24
White blood cell decreased (Investigations) | 12 | 4
Anemia (Blood and lymphatic system disorders) | 3 | 5
Diarrhea (Gastrointestinal disorders) | 3 | 4
Lymphocyte count decreased (Investigations) | 6 | 1
Nausea (Gastrointestinal disorders) | 2 | 5
Fatigue (General disorders) | 2 | 3
Hypertension (Vascular disorders) | 1 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Platelet count decreased (Investigations) | 2 | 1
Sepsis (Infections and infestations) | 1 | 2
Alanine aminotransferase increased (Investigations) | 2 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Blurred vision (Eye disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Joint infection (Infections and infestations) | 1 | 0
Nervous system disorders (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Typhlitis (Gastrointestinal disorders) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Shingles (Infections and infestations) | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Optic nerve disorder (Eye disorders) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sacituzumab Govitecan + Pembrolizumab (N=52) | Sacituzumab Govitecan (N=52)
Neutrophil count decreased (Investigations) | 8 | 8
White blood cell decreased (Investigations) | 3 | 4
Anemia (Blood and lymphatic system disorders) | 15 | 10
Diarrhea (Gastrointestinal disorders) | 9 | 16
Lymphocyte count decreased (Investigations) | 3 | 2
Nausea (Gastrointestinal disorders) | 14 | 12
Fatigue (General disorders) | 18 | 15
Hypertension (Vascular disorders) | 4 | 1
Platelet count decreased (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2
Alkaline phosphatase increased (Investigations) | 7 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 20
Anorexia (Metabolism and nutrition disorders) | 6 | 9
Constipation (Gastrointestinal disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 2 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1
Hypothyroidism (Endocrine disorders) | 3 | 0
Infections and infestations (Infections and infestations) | 4 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0
Insomnia (Psychiatric disorders) | 6 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pain (General disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sinusitis (Infections and infestations) | 1 | 3
Upper respiratory infection (Infections and infestations) | 3 | 6
Urinary tract infection (Infections and infestations) | 3 | 3
Dysgeusia (Nervous system disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT04448886/Prot_SAP_000.pdf